CLINICAL TRIAL: NCT00696813
Title: PILAR: Pharmacoepidemiologic International Longitudinal Antipsychotic Registry
Brief Title: Observational Study to Assess Outcomes During Antipsychotic Treatment With Paliperidone ER or Other Oral Antipsychotics
Acronym: PILAR
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: EMEA Therapeutic Area Leader CNS, Janssen-Cilag Germany
Other Study IDs: CR014707; R076477SCH4016 (Other: Janssen-Cilag International NV); NCT01615133 (obsolete NCT alias)
Record Dates: First submitted 2008-06-05; First posted 2008-06-13 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: Registry; Healthcare Utilization; Outcome; Safety; Efficacy; Cost-effectiveness; Paliperidone ER; Invega®; Oral antipsychotics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- paliperidone ER: Newly switched to or started on Paliperidone ER, not longer than 2 weeks ago
- Any other oral antipsychotic: Newly switched to or started on any other oral antipsychotic treatment (either atypical or conventional), not longer than 2 weeks ago

SUMMARY:
The purpose of this non-interventional, observational and international registry study is to document the prescribing patterns in daily clinical practice and to assess long term treatment outcomes related to initiation of treatment with oral antipsychotics in a naturalistic setting.

DETAILED DESCRIPTION:
PILAR is a non-interventional, observational, international registry on the use of oral antipsychotics in a naturalistic setting in patients with schizophrenia. Patients initiating a new oral antipsychotic treatment are candidates for documentation in this registry. All patients should be treated according to local labeling specifications. The overall study objective is to document prescribing patterns in daily clinical practice and to assess long-term treatment outcomes related to initiation of treatment with oral antipsychotics in a naturalistic setting. The primary objective is to prospectively document over one year treatment outcomes and healthcare utilization data that will enable a cost-effectiveness analysis of paliperidone ER compared to other oral antipsychotic treatments. Additional objectives are to retrospectively collect data over one year, which will allow the evaluation of treatment outcomes before and after treatment initiation with paliperidone ER or other oral antipsychotics. Evaluation of Adverse Drug Reactions (ADR) and Serious Adverse Drug Reactions (SADR) for the retrospective period, and Adverse Events (AE) and Serious Adverse Events (SAE) during the prospective period will be performed and reported. Dosing and administration of all treatments should be prescribed at the physician's discretion, and should be based on approved local labels. Dose adjustments or medication changes should be made by the treating physician based on clinical judgment and usual practice. Subjects should receive their medication according to usual care in their treatment setting, and no study drug will be provided. The documentation of the treatment will last one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Switch to or start on paliperidone ER or another oral antipsychotic treatment (either atypical or conventional), not longer than 2 weeks ago
* Signed informed consent is available at the beginning of documentation
* Able and willing to fill-out self-administered questionnaires

Exclusion Criteria:

* Established treatment-refractory schizophrenia
* History of neuroleptic malignant syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of medical health professionals with a diagnosis of schizophrenia
Sampling Method: Probability Sample
Enrollment: 3064 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Primary treatment duration and time to treatment discontinuation | Prospective 1-year observation period
  Primary treatment duration is defined as the time interval (in days) between baseline and stop of the new antipsychotic treatment started at baseline.

SECONDARY OUTCOMES:
The prospectively documented treatment outcomes also include overall severity of symptoms, personal and social performance, healthcare utilization and health related quality of life and quality of sleep. | 12 months
Use of concomitant medications | during a retrospective period of 3 months and at month 3, 6, 9 and 12 after baseline or early discontinuation
  Use (Yes/No) of each class of concomitant medications
Deterioration of the psychotic condition | at baseline and at month 3, 6, 9 and 12 after baseline or early discontinuation
  A significant deterioration of the psychotic condition is defined as 1 of the following: (a) full hospitalization for exacerbation of psychotic symptoms, (b) need for an increase in level of care, antipsychotic dose increase other than for titration, change in concomitant medication to treat the psychotic symptoms combined with a worsening of psychotic symptoms equivalent to an increase in CGI-S by at least 2 points, (c) deliberate self-injury, (d) emergence of suicidal or homicidal ideation, (e) violent behavior resulting in significant injury to another person or significant property damage

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (84):
- Canada (10):
  - Victoria, British Columbia
  - Burlington, Ontario
  - Chatham, Ontario
  - Greater Sudbury, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Montreal, Quebec
  - Halifax
  - London
  - Windsor
- Czechia (32):
  - Boskovice
  - Brno
  - Brno - Lesná
  - Brno-Židenice
  - České Budějovice
  - Český Krumlov
  - Děčín
  - Frýdek-Místek
  - Hradec Králové
  - Jindřichův Hradec
  - Kolín
  - Kutná Hora
  - Litoměřice
  - Litomyšl
  - Lnáře
  - Mladá Boleslav
  - Nový Jičín
  - Olomouc
  - Ostrava
  - Ostrava-Poruba
  - Pardubice
  - Pilsen
  - Písek
  - Prague
  - Přerov
  - Roudnice
  - Sternberk
  - Teplice
  - Třebíč
  - Ústí nad Labem
  - Vyškov
  - Zábřeh
- Denmark (8):
  - Aarhus C
  - Augustenborg
  - Copenhagen
  - Frederiksberg
  - Gentofte Municipality
  - Middelfart
  - Odense C
  - Toender
- Kazakhstan (5):
  - Almaty
  - Astana
  - Petropavlovsc
  - Shymkent
  - Taldykorgan
- Sweden (16):
  - Borås
  - Bromma
  - Falköping
  - Falun
  - Gothenburg
  - Härnösand
  - Jönköping
  - Ljungby
  - Malmo
  - Mölndal
  - Norrköping
  - Sundsvall
  - Tyresö
  - Uddevalla
  - Varberg
  - Västra Frölunda
- Thailand (2):
  - Khon Kaen
  - Songkhla
- Ukraine (11):
  - Berehove
  - Donetsk
  - Hlevakha
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kryvyi Rih
  - Simferopol
  - Smila
  - Uzhhorod
  - Vinnitsa

REFERENCES:
- [Derived] Schreiner A, Hargarter L, Hitschfield K, Lee JI, Lenskaya I, Sulaiman AH, Diels J; PILAR study group. Clinical effectiveness and resource utilization of paliperidone ER for schizophrenia: Pharmacoepidemiologic International Longitudinal Antipsychotic Registry (PILAR). Curr Med Res Opin. 2014 Jul;30(7):1279-89. doi: 10.1185/03007995.2014.898630. Epub 2014 Mar 19. PMID 24597755
- See also: Pharmacoepidemiologic International Longitudinal Antipsychotic Registry PILAR — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=397&filename=CR014707_CSR.pdf